CLINICAL TRIAL: NCT00100711
Title: Phase II Trial of Motexafin Gadolinium (MGd) in Patients With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma With Refractory or Relapsed Disease
Brief Title: Study of Motexafin Gadolinium (MGd) in Patients With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0222
Record Dates: First submitted 2005-01-04; First posted 2005-01-05 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Leukemia; Lymphoma; Motexafin Gadolinium; Relapsed Chronic Lymphocytic Leukemia; Relapsed Chronic Lymphocycic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Lymphoma | interventions — motexafin gadolinium

INTERVENTIONS:
Drug: Motexafin Gadolinium

SUMMARY:
The primary purpose of this study is to determine if motexafin gadolinium may be an effective treatment for patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL). Secondly, the duration of response and the time during which patients survive without chronic lymphocytic leukemia or small lymphocytic lymphoma worsening will be evaluated. Additionally, the patient's response to motexafin gadolinium will be compared to the response of the patient's cells in a laboratory to motexafin gadolinium.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* CLL as defined by the NCI 96 criteria (exception; patients may have bright surface immunoglobulin staining if negative for t[11;14] translocation or cyclin D1) or SLL as defined by WHO classification criteria and is refractory or relapsed as defined by one of the following: 1) Refractory disease- progressive disease while on therapy, or 2) Relapsed disease progressive disease after at least one treatment course of therapy with disease response or stabilization
* ECOG performance status score of 0, 1, or 2
* Willing and able to provide written informed consent

Exclusion Criteria:

Laboratory Values of:

* Platelet count < 30,000/µL
* AST or ALT > 2 x ULN (upper limit of normal)
* Total bilirubin > 2 x ULN
* Creatinine > 2.0 mg/dL

and

* Chemotherapy, radiation therapy, immunotherapy, systemic corticosteroids (> 10 mg oral prednisone or equivalent), or systemic biologic anticancer therapy within 21 days before beginning study treatment
* Greater than three prior regimens (where a regimen is defined as a treatment for CLL/SLL given initially or after disease progression)
* Uncontrolled hypertension
* Known history of porphyria (testing not required at screening)
* Known history of glucose-6-phosphate dehydrogenase (G6PD) deficiency (testing not required at screening)
* Known history of HIV infection (testing not required at screening)
* Pregnant or lactating (pregnancy test is required for all female patients of childbearing potential)
* Woman of childbearing potential or sexually active man unwilling to use adequate contraceptive protection
* Physical or mental condition that makes patient unable to complete specified follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27
Dates: Start 2004-10; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Complete and partial response rates

SECONDARY OUTCOMES:
Progression-free survival
Duration of response
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Evens, D.O., Principal Investigator — Robert H. Lurie Comprehensive Cancer Center of Northwestern University; Neil E. Kay, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - The Mayo Clinic, Rochester, Minnesota
  - The Ohio State University, Columbus, Ohio